CLINICAL TRIAL: NCT01079338
Title: Salivary Proteome and Sensitivity to Bitterness
Acronym: PROTAMER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Purpose: Basic Science
Other Study IDs: AFSSAPS-2009-A00320-57
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2010-03-03 (Estimated); Status verified 2010-02

CONDITIONS: Healthy
Keywords: sensitivity to caffeine
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- caffeine (Experimental)
  Interventions: Other: caffeine

INTERVENTIONS:
Other: caffeine

SUMMARY:
This study aims to establish whether the protein composition of healthy males contribute to their sensitivity to the bitterness of caffeine.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* smokers
* currently suffering from oral pathologies
* sensory aversion to bitterness

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Martine Morzel, PhD, Principal Investigator — Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement